CLINICAL TRIAL: NCT06469125
Title: Multicentric Prospective Evaluation of Bladder Injuries During Morcellation Using BICEP (Bladder Injury Classification During Endoscopic Procedures)
Brief Title: Anatomic Endoscopic Prostate Enucleation and BICEP Classification
Acronym: BICEP
Status: Completed | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Collaborators: Danube University Krems (Other); University General Hospital of Heraklion (Other); Paracelsus Medical University (Other); University of Turin, Italy (Other); Menoufia University (Other); Acibadem Ankara Hospital (Other); Universitätsmedizin Mannheim (Other); Martini-Klinik am UKE GmbH (Other); Asklepios Kliniken Hamburg GmbH (Other); Istanbul Medipol University Hospital (Other); Saint Petersburg State University, Russia (Other); HM Sanchinarro University Hospital (Other); Alexandria University (Other); Spital Thurgau AG (Other); Medical University of Graz (Other); King's College Hospital NHS Trust (Other); Sheikh Khalifa Medical City (Other)
Responsible Party: Principal Investigator, Selim Soyturk, Research Assistant, Necmettin Erbakan University
Other Study IDs: ResCORE-2024-12
Record Dates: First submitted 2024-06-04; First posted 2024-06-21 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-05

CONDITIONS: Bladder Injury; Prostate Hyperplasia
Keywords: BICEP classification; Anatomic Endoscopic Enucleation of Prostate; Bladder Injury; HoLEP; BiLEP; ThuFLEP
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Morcellation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic Prostate Interventions for Anatomic Enucleation — The intervention in this study involves performing anatomic endoscopic enucleation of the prostate (AEEP) using different energy sources. Following the enucleation, the resected prostate tissue will be morcellated within the bladder using various morcellators to remove the enlarged prostate tissue minimally invasively. The process will also involve evaluating and categorizing any resulting bladder injuries using the BICEP classification system.
  Other Names: Morcellation

SUMMARY:
The Bladder Injury Classification System for Endoscopic Procedure (BICEP) is designed to provide a systematic framework for categorizing bladder injuries that occur during endoscopic procedures. By standardizing the classification of these injuries, BICEP promotes a more consistent approach to diagnosis, management, and prevention across different urologic interventions. This study aims to validate and implement the BICEP system during morcellation.

This study will:

Validate BICEP by using real-life clinical scenarios to ensure its applicability and effectiveness.

Assess the incidence and types of bladder injuries during morcellation, using the BICEP categorization to standardize injury reporting and enhance treatment protocols.

DETAILED DESCRIPTION:
Insufficient knowledge exists about bladder injuries during morcellation, as the existing literature primarily consists of isolated case reports. The Bladder Injury Classification System for Endoscopic Procedures (BICEP) aims to standardize the reporting and management of bladder injuries during endoscopic surgeries.

This study proposes an external validation of the BICEP system through an international, multicenter, prospective observational study. The objectives of this study are fourfold:

Validate the newly developed BICEP classification system with real-life clinical scenarios to ensure its applicability and effectiveness.

Evaluate the incidence and types of bladder injuries during morcellation using the BICEP framework to standardize injury reporting and enhance treatment protocols.

Assess the robustness of BICEP across different departments. Facilitate the adoption of BICEP as a global standard for classifying bladder injuries in endoscopic surgery.

Through this study, the validity of BICEP will be confirmed and the bladder injuries occurring during morcellation after AEEP will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥40
* ASA (American Society of Anesthesiologists) score ≤4
* Patients undergoing Holmium Laser Enucleation of the Prostate (HoLEP) or Transurethral Resection of the Prostate (TURP) surgery.

Exclusion Criteria:

* Patients with neurological disorders that may affect bladder function, such as cerebrovascular stroke or Parkinson's disease.
* Patients with active urinary tract infection.
* Patients diagnosed with bladder cancer within the last 2 years.
* Patients with prostate cancer.
* Patients who have undergone previous prostate surgery.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will include adult patients undergoing AEEP surgery. The presence of bladder injuries during the operation will be assessed according to the BICEP classification, and any potential injuries will be recorded.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2025-10-08 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Successful Validation of the Bladder Injury Classification System for Endoscopic Procedure Classification System for Bladder Injuries Occurring During Morcellation in AEEP Operations | Up to 24 weeks
  Approximately 250 participants will be evaluated using a scoring system ranging from 0 to 4 to assess the severity of the injury. A score of 0 indicates no injury, while a score of 4 indicates extensive avulsion of part of the bladder. In this system, the severity of the injury increases as the score increases.
The impact of different energy sources and morcellation devices on bladder injury | Up to 24 weeks
  The severity of the injury will be assessed using a scoring system ranging from 0 to 4. A score of 0 indicates no injury, while a score of 4 indicates the highest degree of avulsion of part of the bladder. In this system, the severity of the injury increases as the score increases.

SECONDARY OUTCOMES:
Postoperative Qmax Increase Following Morcellation in AEEP Operations | 1 month post surgery
  Assessed by maximum flow rate (Q-max) measured using uroflowmetry by ml/sec, better outcome above 15ml/sec
Postoperative Improvement in International Prostate Symptom Score (IPSS) | 1 month post surgery
  The IPSS form will be filled out for calculation. Scores of 0-7 indicate mild symptoms, 8-19 indicate moderate symptoms, and 20-35 indicate severe symptoms.
Duration of catheterization | Up to 10 weeks
  The duration of catheterization post-operation will be calculated in days.
Length of hospital stay | Up to 6 weeks
  The duration of hospital stay post-operation will be calculated in days.

CONTACTS AND LOCATIONS:
Overall Officials: Selçuk Güven, Prof. Dr., Study Director — Necmettin Erbakan University; Bülent Erkurt, Prof. Dr., Study Chair — Istanbul Medipol University Hospital; Selim Soytürk, RA, Principal Investigator — Necmettin Erbakan University
Locations (2):
- Turkey (Türkiye) (2):
  - Necmettin Erbakan University, Konya, Konya
  - Istanbul Medipol University Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Result] Breda A, Gallioli A, Diana P, Fontana M, Territo A, Gaya JM, Rodriguez-Faba O, Huguet J, Piana A, Verri P, Baboudjian M, Aumatell J, Algaba F, Palou J. The DEpth of Endoscopic Perforation scale to assess intraoperative perforations during transurethral resection of bladder tumor: subgroup analysis of a randomized controlled trial. World J Urol. 2023 Oct;41(10):2583-2589. doi: 10.1007/s00345-022-04052-w. Epub 2022 Jun 4. PMID 35665840
- [Result] Gilling PJ, Kennett K, Das AK, Thompson D, Fraundorfer MR. Holmium laser enucleation of the prostate (HoLEP) combined with transurethral tissue morcellation: an update on the early clinical experience. J Endourol. 1998 Oct;12(5):457-9. doi: 10.1089/end.1998.12.457. PMID 9847070
- See also: A case of blunt abdominal trauma resulting in significant bladder injury (AAST grade IV) — https://www.ijcriurology.com/archive/2022/pdf/100027Z15DB2022.pdf